CLINICAL TRIAL: NCT04962711
Title: Risk-guided Disease Management Plan to Prevent Heart Failure in Patients Treated With Previous Chemotherapy (REDEEM)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baker Heart and Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 82/21
Record Dates: First submitted 2021-06-22; First posted 2021-07-15 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Randomization to CO-DMP or usual care
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will receive study data based on pooled de identified dataset.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heart failure intervention ( Cardio-Oncology Disease Management Plan (CO-DMP) (Experimental): 1. Optimization of pharmacotherapy: Cardioprotection with angiotensin-converting enzyme inhibitor (ACEi, Ramipril) and beta blocker (Metoprolol).Participants will be initially treated with ramipril at a dose of 1.25 or 2.5mg (according to baseline systemic arterial pressure), once or twice a day, and gradually up-titrated to 10mg/day, or to the maximal-tolerated dose. In patients receiving at least 2.5mg/day of ramipril, metoprolol will be started at an initial dose of 50 (25mg twice a day) and progressively up-titrated to the maximal dose of 100mg/day. Patients will be reviewed every 2 weeks during the up titration phase.
  2. Exercise intervention: Individualized training program provided by an exercise physiologist.
  Interventions: Other: Heart Failure intervention (Cardio-Oncology Disease Management Plan (CO-DMP)
- Usual care (Active Comparator): Provided by participants' usual healthcare professional(s), guided by a brochure regarding optimal risk factor management addressing hypertension, lipids, alcohol intake and tobacco use.
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Heart Failure intervention (Cardio-Oncology Disease Management Plan (CO-DMP) — A clinical review to ensure optimal risk factor control and cardioprotection along with exercise intervention.
  Arms: Heart failure intervention ( Cardio-Oncology Disease Management Plan (CO-DMP)
Other: Usual care — provided by participants' usual healthcare professional(s)
  Arms: Usual care

SUMMARY:
This is a prospective study in which a process of identifying and reducing heart failure (HF) risk will be applied to cancer survivors >55 years old with chemotherapy >5 years ago.

The overall goal of this study to identify the feasibility and value of risk-guided cardiac rehabilitation (exercise, risk factor modification, and behavioural support) as a component of survivorship care.

DETAILED DESCRIPTION:
Participants enrolled in this study will be randomized to cardio-oncology disease management plan ( CO-DMP) that involves the use of surveillance imaging to detect subclinical left ventricular dysfunction (LVD), clinical review to ensure optimal risk factor control and cardio-protection and exercise/sedentariness intervention. The intervention will be delivered over a period of 6 months. Usual care patients will then cross over the CO-DMP for 6 months. The outcome from this study will show that subclinical LVD is more common among long term cancer survivors, and a CO-DMP is feasible in reducing HF risk factors in this sub group of survivors.

ELIGIBILITY:
Inclusion Criteria:

1. History of cancer > 10 years ago
2. Have received potentially toxic chemotherapy Anthracycline (any dose) Trastuzumab (Herceptin) in breast-cancer with the HER2 mutation OR Tyrosine kinase inhibitors (e.g. sunitinib) OR Left chest radiotherapy

Exclusion Criteria:

1. Ejection fraction at baseline echo <50%
2. Valvular stenosis or regurgitation of >moderate severity
3. History of previous heart failure (baseline New York Heart Association (NYHA) classification >2)
4. Systolic BP <110 mmHg
5. Pulse <60/minute if not on beta blocker
6. Inability to acquire interpretable images (identified from baseline echo)
7. Contraindications to beta blockers or angiotensin-converting enzyme inhibitors
8. Oncologic (or other) life expectancy <12 months or any other medical condition (including pregnancy) that results in the belief (deemed by the Chief Investigators) that it is not appropriate for the patient to participate in this trial
9. Already taking both angiotensin converting enzyme inhibitors/angiotensin receptor blockers and beta blockers, or intolerance (or allergy) to both.
10. Unable to provide written informed consent to participate in this study

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 685 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in exercise capacity | Over a period of 6 months
  Cardio pulmonary fitness (peak oxygen uptake (VO2 peak)) from baseline to follow up.

SECONDARY OUTCOMES:
Medication adherence | Over a period of 6 months
  proportion of ACEi and beta blocker tablets taken
Neuromuscular strength | Over a period of 6 months
  Maximal isometric grip strength (kg) assessed using a digital grip strength dynamometer
Endurance | Over a period of 6 months
  Increase in total exercise duration.
Left ventricular function | Over a period of 6 months
  Change in global longitudinal strain (GLS) using echocardiographic speckle-tracking

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Marwick, MD,PhD,MPH, Principal Investigator — Baker Heart and Diabetes Institute
Locations (1):
- Baker Heart and Diabetes Institute, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No
Data sharing based available on application to the study PI

REFERENCES:
- [Derived] Wong J, Smith J, Soh CH, Howden E, Talbot JS, Nolan M, Whitmore K, Wright L, Sherriff AG, Sivaraj E, Wheeler G, Wiltshire K, Campbell P, Ramkumar S, Tam C, Marwick TH. Risk-guided disease management to prevent heart failure in adult cancer survivors of previous cardiotoxic cancer treatments: Baseline results of the REDEEM trial. Am Heart J. 2026 Feb;292:107277. doi: 10.1016/j.ahj.2025.09.009. Epub 2025 Sep 16. PMID 40967296